CLINICAL TRIAL: NCT06191081
Title: Intraoperative Identification of the Optimal Functional Lymphatic Vessel for Lymphaticovenous Anastomosis in Upper Limb Extremity Lymphedema
Brief Title: Identification of the Optimal Functional Lymphatic Vessel for Lymphaticovenous Anastomosis
Status: Completed | Type: Observational
Sponsor: Taizhou Hospital (Other)
Responsible Party: Principal Investigator, Haihua Yang, Chief Physician, Taizhou Hospital
Other Study IDs: FLV20231208
Record Dates: First submitted 2023-12-10; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Lymphedema
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: lymphaticovenous anastomosis — lymphaticovenous anastomosis

SUMMARY:
The aim of this study is to further explore the optimal screening factors for functional lymphatic vessels in lymphaticovenous anastomosis in patients with lymphedema.

DETAILED DESCRIPTION:
By analyzing the size of lymphatic vessels (0.3-0.6mm), ICG imaging, contraction characteristics of lymphatic vessels and lymphatic flow in patients with lymphedema, the effect of functional lymphatic vessel selection on lymphatic drainage in patients with lymphedema was judged during operation, so as to provide a more scientific basis for the selection of functional lymphatic vessels in clinical surgery.

ELIGIBILITY:
Inclusion Criteria:

* lymphedema Paitent

Exclusion Criteria:

* myoedema Paitent；lipedema Paitent

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Aged 18-80 years; Lymphedema and swelling of the limbs for more than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Rate of size(0.3-0.6mm) | through study completion, an average of 2.5 year
  size of lymphatic vessels
Rate of lymphatic vessels contractility | through study completion, an average of 2.5 year
  When observing lymphatic vessels in fluorescence mode, a contraction occurring within 10 seconds is considered as contractility positive
Rate of flow | through study completion, an average of 2.5 year
  while the presence of lymphatic fluid flowing out after cutting the lymphatic vessel is considered as flow positive
Rate of ICG | through study completion, an average of 2.5 year
  When observing lymphatic vessels in fluorescence mode, lymphatic vessel fluorescence is considered as ICG positive

CONTACTS AND LOCATIONS:
Overall Officials: youmao liu, Study Director — employee
Locations (1):
- Chong Liu, Zhejiang, China